CLINICAL TRIAL: NCT06753409
Title: Impact of Reduced Intraoperative Norepinephrine Requirements Via Processed Electroencephalography-Guided General Anesthesia on Patient Outcomes After Major Abdominal Surgeries
Brief Title: Processed Electroencephalography-guided General Anesthesia and Outcomes in Major Abdominal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, walaa hamdy mohamed hemaid, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EEG-Guided General Anesthesia
Record Dates: First submitted 2024-12-10; First posted 2024-12-31 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Acute Kidney Injury
Keywords: Hypotension; Abdominal surgery; Norepinephrine; Acute kidney injury
MeSH Terms: conditions — Hypotension; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pEEG-Guided General Anesthesia Group (Active Comparator): Depth of anesthesia will be managed based on pEEG monitoring using Entropy with a target range of 40-60.
  Interventions: Device: Processed electroencephalography (pEEG) Guided General Anesthesia
- Non-pEEG-Guided Anesthesia (Standard Care Group) with blinded pEEG monitoring (Placebo Comparator): Depth of anesthesia will be managed based on clinical judgment, informed by clinical perception and vital signs.
  Interventions: Device: Non-pEEG-Guided General Anesthesia (with blinded pEEG monitoring)

INTERVENTIONS:
Device: Processed electroencephalography (pEEG) Guided General Anesthesia — Processed electroencephalography (pEEG) can guide the optimization of anesthesia depth, potentially preventing overly deep anesthesia and, in turn, reducing the incidence of IOH and the need for vasopressors .
  Depth of anesthesia will be managed based on pEEG monitoring using Entropy with a target range of 40-60.
  Arms: pEEG-Guided General Anesthesia Group
Device: Non-pEEG-Guided General Anesthesia (with blinded pEEG monitoring) — Depth of anesthesia will be managed based on clinical judgment, informed by clinical perception and vital signs.
  Arms: Non-pEEG-Guided Anesthesia (Standard Care Group) with blinded pEEG monitoring

SUMMARY:
This study aims to evaluate whether the reduction in the amount of intraoperative norepinephrine required to prevent hypotension, facilitated by processed electroencephalography (pEEG) -guided general anesthesia, will lead to a decrease in postoperative complications, particularly acute kidney injury (AKI).

DETAILED DESCRIPTION:
In major abdominal surgery, intraoperative hypotension (IOH) remains a prevalent concern, contributing significantly to postoperative complications. These complications include acute kidney injury (AKI), myocardial injury, and even mortality. While IOH is multifactorial, its occurrence is frequently associated with the need for vasopressor support, particularly norepinephrine, which is widely used to manage and prevent IOH. However, it is important to note that vasopressors, including norepinephrine, are themselves implicated in promoting AKI .

The lack of consensus on a universal definition for IOH adds complexity to this issue. Currently, it remains unclear whether IOH should be defined based on absolute blood pressure thresholds or as a relative decrease from baseline. IOH is commonly defined as a systolic blood pressure of <90 mm Hg or a mean arterial pressure (MAP) of <65 mm Hg.

Ephedrine is often the first-line vasopressor administered to treat IOH, with norepinephrine as a second-line option. The hemodynamic effects of these two agents differ: norepinephrine increases cardiac preload without significantly increasing afterload, thereby raising cardiac output. Ephedrine, however, increases cardiac output but with a greater increase in afterload, often leading to tachycardia, which can be detrimental to patients. The variable effectiveness of ephedrine and its associated side effects have led clinicians to consider norepinephrine as a more appropriate option for managing IOH, potentially with fewer cardiovascular side effects.

Additionally, crystalloid fluid overload during abdominal surgery has been linked to poor postoperative outcomes, including anastomotic instability. Liberal fluid regimes may disrupt the physiological healing processes at surgical sites, suggesting that fluid management strategies aimed at minimizing overload could improve patient outcomes.

Recent studies propose that early norepinephrine administration to maintain MAP, even before the onset of hypotension, may help reduce the need for large fluid volumes.

One important factor contributing to IOH and vasopressor use is excessively deep general anesthesia. Processed electroencephalography (pEEG) can guide the optimization of anesthesia depth, potentially preventing overly deep anesthesia and, in turn, reducing the incidence of IOH and the need for vasopressor .

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for major abdominal surgery lasting more than 2 hours under general anesthesia.
2. American Society of Anesthesiologists Physical Status (ASA) score I-III.
3. Age range of 18-70 years.
4. Both male and female patients.

Exclusion Criteria:

1. Emergency surgeries.
2. Uncontrolled hypertension (systolic blood pressure >150 mm Hg) despite medication.
3. Recent acute cardiovascular events, including heart failure or acute coronary syndrome.
4. Chronic kidney disease with a glomerular filtration rate <30 ml/min/1.73 m² or requiring renal replacement therapy.
5. Severe hepatic failure (ASAT/ALAT >2N, elevated bilirubin, or PT <50%).
6. Preoperative sepsis or septic shock.
7. Pregnancy.
8. Patient refusal to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative acute kidney injury (AKI) based on the KDIGO criteria. | Assessed at the third postoperative day.
  Diagnosis and severity of PO-AKI will be assessed by serum-creatinine and/or urine output according to the KDIGO criteria .
  The latest serum creatinine before surgery will be defined as baseline value. Serum creatinine will be measured at least once a day for the first 3 days. Patients with serum creatinine increases of ≥0.3 mg/dl within 48 h or 1.5-1.9 times increases within 72 h after surgery will be diagnosed KDIGO stage 1, patients with serum creatinine increases of 2-2.9 times within 72 h will be diagnosed KDIGO stage 2, and patients with serum creatinine increases of ≥3 times or ≥4 mg/dl or with the need of renal replacement therapy (RRT) will be diagnosed KDIGO stage 3.
  Further, patients with a urine out- put <0.5 ml/kg/h for ≥6 h will be diagnosed KDIGO stage 1, urine output <0.5 ml/kg/h for ≥12 h KDIGO stage 2, and <0.3 ml/kg/h for ≥24 h or anuria for ≥12 h KDIGO stage 3. Once the urine catheter removed, the urine output criterion will no longer be considered.

SECONDARY OUTCOMES:
1.Total dose of norepinephrine administrated | 48 hour
  The total cumulative dose of norepinephrine administered intraoperatively and postoperatively will be recorded in micrograms.
2.The volume of intraoperative fluid therapy. | 48 hour
  The volume of crystalloids, colloids, and blood products administered intraoperatively will be recorded in (milliliters).

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No